CLINICAL TRIAL: NCT06284109
Title: Preoperative (Pre-amputation) Cryoanalgesia to Improve Post-amputation Phantom Limb Pain, General Physical and Emotional Disability, and Opioid Consumption: a Randomized Pilot Trial
Brief Title: Preoperative (Pre-amputation) Cryoanalgesia to Improve Post-amputation Phantom Limb Pain
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment challenges
Sponsor: The Cleveland Clinic (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23-1036
Record Dates: First submitted 2024-01-30; First posted 2024-02-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative Pain; Phantom limb syndrome; Postoperative movilization; Lower limb amputation
MeSH Terms: conditions — Pain, Postoperative; Phantom Limb

STUDY DESIGN:
Intervention Model Description: Pre-Operative Patients will receive cryoanalgesia or sham cryoanalgesia before amputation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All participants will receive nerve blocks with Local anesthetic. Participants will be Randomized on a 1:1 fashion to cryoanalgesia or sham cryoanalgesia, based on computer-generated codes and use random-sized blocks. Patients will not be told which group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cryoanalgesia (Experimental): Participants will receive cryoanalgesia with the The iovera° system.
  Interventions: Device: Cryoanalgesia
- Sham Cryoanalgesia (Sham Comparator): Participants will receive Sham cryoanalgesia with the The iovera° system.
  Interventions: Device: Sham Cryoanalgesia

INTERVENTIONS:
Device: Cryoanalgesia — Participants will receive cryoanalgesia with the The iovera° system. . The specific nerves targeted will be both the sciatic, targeted first (as distal as possible, but not more distal than the bifurcation), and femoral, targeted second (as distal as possible, but not more distal than the adductor canal). Cryoanalgesia will result from an 8-minute-long percutaneous cryoneuroablation procedure consisting of several freeze/defrost cycles. Per routine, all patients will have a nerve block with single shot ropivacaine.
  Arms: Cryoanalgesia
Device: Sham Cryoanalgesia — Participants will receive Sham cryoanalgesia with the The iovera° system. The specific nerves targeted will be both the sciatic, targeted first (as distal as possible, but not more distal than the bifurcation), and femoral, targeted second (as distal as possible, but not more distal than the adductor canal). Per routine, all patients will have a nerve block with single shot ropivacaine.
  Arms: Sham Cryoanalgesia

SUMMARY:
Investigators will evaluate preamputation cryoanalgesia on pain, mobility, opioid use and general physical and emotional disability using a pilot randomized trial design, to explore the amount and variability of improvement on those outcomes and to investigate the potentiality of conducting a future larger randomized controlled trial, which the investigators will assess quantitatively the benefits of cryoanalgesia.

DETAILED DESCRIPTION:
Primary Aim: To determine preoperative cryoneurolysis improves phantom limb pain compared with no cryoneurolysis. Estimate the standard deviation of phantom limb pain score at baseline and post-treatment (Day 0), Days 1 and 2; Weeks 1, 2, 3, and Months 1, 2 and 3. The investigators will consider using the upper limit of the 75% confidence interval to plan the sample size of future larger trial.

Hypothesis 1: Preoperative cryoneurolysis reduces phantom limb pain over 3 month after surgical leg amputation compared with no cryoneurolysis.

Secondary Aim 1: To determine if preoperative cryoneurolysis improves mobility after lower limb amputation compared with no cryoneurolysis.

Hypothesis 1: Preoperative cryoneurolysis improves mobilization (as measured with accelerometer) over 3 the month after surgical leg amputation compared with no cryoneurolysis.

Secondary Aim 2: To determine if preoperative cryoneurolysis improves general physical and emotional disability after lower limb amputation compared with no cryoneurolysis.

Hypothesis 2: Preoperative cryoneurolysis reduces general physical and emotional disability (as measured with the World Health Organization Disability Assessment) over the 3 month after surgical leg amputation compared with no cryoneurolysis.

Secondary Aim 3: To determine if preoperative cryoneurolysis decreases opioid use after lower limb amputation compared with no cryoneurolysis.

Hypothesis 3: Preoperative cryoneurolysis reduces opioid consumption over the 3 month after surgical leg amputation compared with no cryoneurolysis.

Exploratory Aims:

Hypothesis 1: Preoperative cryoneurolysis reduces residual limb pain over the 3 months after surgical leg amputation compared with no cryoneurolysis.

ELIGIBILITY:
Inclusion Criteria:

* Adults at least 18 years of age.
* Scheduled for a unilateral lower limb amputation distal to the femoral head and including at least one metatarsal bone.

Exclusion Criteria:

* Pregnancy
* Incarceration
* Morbid obesity (body mass index greater than 40 kg/m2
* Contraindication specific to cryoneurolysis such as a localized infection at the treatment site, cryoglobulinemia, cold urticaria, or Reynaud's syndrome.
* Investigator opinion that the potential subject is a poor candidate for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Phantom limb pain score | 3 Months
  Pain scores ranging from 0 - "no pain" to 10 - "worst pain ever" over 3 month after surgical leg amputation.

SECONDARY OUTCOMES:
Mobility | 3 Months
  Number of steps measured with accelerometer integrated into the Fitbit Inspire 3 Health &-Fitness-Tracker) over 3 the month after surgical leg amputation compared with no cryoneurolysis.
General physical and emotional disability | 3 Months
  General physical and emotional disability measured with the World Health Organization Disability Assessment. Level of disability is described as none (0-0.49), mild (0.5-1.49), moderate (1.5-2.49), severe (2.5-3.49), or extreme (3.5-4).
Opioid consumption | 3 Months
  Opioid consumption measured by Morphine Equivalent Doses over 3 months after surgical leg amputation.

OTHER OUTCOMES:
Residual limb pain | 3 Months
  Pain scores ranging from 0 - "no pain" to 10 - "worst pain ever" over 3 month after surgical leg amputation.

CONTACTS AND LOCATIONS:
Overall Officials: Alparslan Turan, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Foundation, Cleveland, Ohio, United States